CLINICAL TRIAL: NCT04324086
Title: Post Operative Pain After Removal of Calcium Hydroxide With Different Activation Techniques
Brief Title: Effect of Removal of Intracanal Medication on Post Operative Pain
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Minia University (Other)
Responsible Party: Principal Investigator, Shaimaa Nasr El-deen Abd El-gaffar, phD student - Endodontic Department, Minia University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 311
Record Dates: First submitted 2020-03-24; First posted 2020-03-27 (Actual); Last update posted 2020-03-27 (Actual); Status verified 2020-03

CONDITIONS: Effects of the Elements

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Masking Description: double
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- XP-endo Finisher file (Experimental): removal of calcium hydroxide intracanal medication with XP-endo Finisher file
  Interventions: Device: Calcium hydroxide with XP-endo Finisher file
- Irrisafe Ultrasonic tip (Experimental): removal of calcium hydroxide intracanal medication with passive ultrasonic irrigation
  Interventions: Device: Calcium hydroxide with Irrisafe Ultrasonic tip
- side vented needle (Active Comparator): removal of calcium hydroxide intracanal medication with conventional syringe irrigation
  Interventions: Device: Calcium hydroxide with side vented needle

INTERVENTIONS:
Device: Calcium hydroxide with XP-endo Finisher file — XP-endo Finisher files (FKG Dentaire, La Chaux-de-Fonds, Switzerland). file will be used with an endodontic motor X-Smart (Dentsply Sirona, Ballaigues, Switzerland) in removal of calcium hydroxide
  Arms: XP-endo Finisher file
Device: Calcium hydroxide with Irrisafe Ultrasonic tip — passive ultrasonic irrigation (PUI) with an IrriSafe Ultrasonic tips (Acteon,France), which will be driven by an ultrasonic device (Newtron P5, Satelec, Acteongroup, Merignac, France) in reemoval of calcium hydroxide
  Other Names: passive ultrasonic irrigation
  Arms: Irrisafe Ultrasonic tip
Device: Calcium hydroxide with side vented needle — conventional syringe irrigation with side vented needle (prime Dent, India) in removal of calcium hydroxide
  Other Names: conventional syringe irrigation
  Arms: side vented needle

SUMMARY:
Recruited patients with necrotic pulp after application of Calcium hydroxide are assigned to group (XP Endo Finisher file) and group( Passive ultrasonic irrigation) and group (conventional syringe irrigation with side vented needle) to remove intracanal medication and record postoperative pain afterwards.

DETAILED DESCRIPTION:
The investigator will recruit patients who are found eligible to the criteria, Calcium hydroxide will be inserted inside the canals. After 7 days, patients will be randomly assigned to either removal of intracanal medication using, the XP-Endo Finisher file, passive ultrasonic irrigation (PUI) and conventional syringe irrigation with side vented needle.

After the visit, patients will be asked to record post operative pain by Visual Analog Scale)in a given sheet

ELIGIBILITY:
Inclusion Criteria:

* Medically free patients.
* Patient's age between 20-50 years.
* Both sexes.
* Necrotic pulp as indicated by thermal or electric pulp testing.
* No history of previous endodontic treatment of the tooth.
* Enough crown structure for adequate isolation.

Exclusion Criteria:

* Pregnancy or lactation
* Medically compromised patients
* Previous endodontic therapy of the affected tooth.
* Teeth diagnosed with vital pulp.
* Teeth with periodontal pocket more than 3mm deep.
* Teeth with abnormal anatomy or calcified canals.
* Teeth with caries below the bony level (non-restorable tooth).
* Immature teeth with open apices.

Ages: 20 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Estimated)
Dates: Start 2020-04-01 (Estimated); Primary Completion 2020-06-01 (Estimated); Study Completion 2020-10-01 (Estimated)

PRIMARY OUTCOMES:
change in post operative pain (Visual Analogue Scale) | Intrappointment at 4,24,48,72 and 96 hours
  Numerical (0-10)

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of Oral and dental medicine, Minia University, Minya, Egypt

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: ICF, CSR

REFERENCES:
- [Background] Sadaf D, Ahmad MZ. Factors associated with postoperative pain in endodontic therapy. Int J Biomed Sci. 2014 Dec;10(4):243-7. PMID 25598754
- [Background] Singh RD, Khatter R, Bal RK, Bal CS. Intracanal medications versus placebo in reducing postoperative endodontic pain--a double-blind randomized clinical trial. Braz Dent J. 2013;24(1):25-9. doi: 10.1590/0103-6440201302039. PMID 23657409
- [Result] Gondim E Jr, Setzer FC, Dos Carmo CB, Kim S. Postoperative pain after the application of two different irrigation devices in a prospective randomized clinical trial. J Endod. 2010 Aug;36(8):1295-301. doi: 10.1016/j.joen.2010.04.012. Epub 2010 Jun 19. PMID 20647083